CLINICAL TRIAL: NCT03970902
Title: The Effectiveness of an Integrated Osteoporosis Care Programme in Postmenopausal Women With Osteoporosis
Brief Title: Quality of Life in Postmenopausal Women With Osteoporosis
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: EC/2019/0578
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Integrated Care; Complex intervention; Primary care; Quality of Life
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Integrated Osteoporosis Care: Group of formal and informal primary caregivers and non-institutionalized postmenopausal women with osteoporosis in whom a complex patient-tailored intervention is provided.
  Interventions: Other: Integrated Osteoporosis Care
- Care As Usual: Group of formal and informal primary caregivers and non-institutionalized postmenopausal women with osteoporosis receiving care as usual for the management of osteoporosis.
  Interventions: Other: Care As Usual

INTERVENTIONS:
Other: Integrated Osteoporosis Care — Complex intervention in family physicians, primary caregivers, patients, informal caregivers. The intervention has a patient-tailored implementation. Family physicians: postgraduate education on osteoporosis management and integrated care, educational material. Primary care stakeholders (nurses, pharmacists, dietitians, physiotherapists): specialist training on patient-support in osteoporosis management with attention towards self-management support (nurses), treatment adherence and administration (pharmacists), fall risk, weight-bearing exercises, balance training and fear of falling (physiotherapists) and anti-inflammatory nutrition with sufficient calcium, vitamin D and protein intake (dietitians). Patients: patient-tailored complex intervention consisting of: education, support consultation(s)/telephones from an osteoporosis nurse, a pharmacist, a physiotherapist and nutritional a dietitian. Informal caregivers: education on supporting osteoporosis self-management.
  Groups: Integrated Osteoporosis Care
Other: Care As Usual — No intervention Patients receive care as usual from their family physician
  Groups: Care As Usual

SUMMARY:
The researchers will evaluate the effectiveness of a complex intervention composed of multiple actions targeting primary care healthcare workers and postmenopausal women with osteoporosis by means of a quasi-experimental design in the form of a cluster-controlled trial with clustering at family physician level. The study has 2 study arms. In one arm, osteoporosis stakeholders receive a complex intervention (Integrated Osteoporosis Care(IOC)). The second study arm serves as control and receives care as usual.

The complex intervention is composed of

* education and provision of educational material for all stakeholders in primary osteoporosis care (patients, family physicians, nurse-educators, physiotherapists, dietitians, pharmacists and if present patient's informal caregivers)
* patient self-management support by primary care osteoporosis stakeholders
* the construction of a primary care osteoporosis treatment guideline and care pathway Effectiveness will be measured by questionnaires and data from the (Electronic Medical Record)EMR and IMA-database, in patients and family physicians.

Effects measured in family physicians are:

* Identification failure rate
* Percentage of family physicians correctly implementing the osteoporosis treatment guideline
* Proportion of patients treated correctly as stated in the osteoporosis treatment guideline
* Proportion of family physicians correctly registering osteoporosis related information in the EMR
* Intensity of collaborative practices
* Knowledge of osteoporosis management and treatment

Effects measured in patients are:

* Medication Possession Ratio(MPR) (Primary outcome)
* Health literacy
* Self-management efficacy
* Self-reported treatment adherence
* Self-reported nutritional intake
* Intensity of integrated osteoporosis care
* Patient satisfaction with integrated osteoporosis care
* HRQoL
* Functional independence (Activities of Daily Living - ADL)
* Patient resource use The study elapse time is 18 months. Participating family physicians will receive postgraduate education and start to include patients during consultations in their doctor's office. The inclusion period is 6 months, patients eligible for participation are non-institutionalized postmenopausal women with a diagnosis of osteoporosis who are able to give informed consent.

The follow-up period for patients is 12 months. Follow-up period for family physicians is 18 months.

DETAILED DESCRIPTION:
Study design:

A quasi-experimental cluster-controlled trial will be conducted with 2 study arms - intervention vs. control - with clustering at GP-level. The cluster design is imperative because the intervention is implemented within the community, and data will be collected at the physician and patient levels. Trial implementation will last 18 months. GPs will be included prior to the study and will enroll patients during a 6-month period; patients will be followed for 12 months. In the IOC-arm, multiple interventions, representing an integrated approach to postmenopausal osteoporosis (PO) management, are offered for implementation. In the control arm, no intervention will take place and patients will receive CAU. The IOC-programme will be offered within the greater region of Ghent (GRG), GPs and patients from the CAU-group will be located outside this region.

Participants:

Participants will be GPs and their patients. For GPs, the only exclusion criterion will be planned retirement during the study period. For GPs in the IOC-arm, willingness to adhere to the newly developed PO management guideline is an extra inclusion criterion. In both arms, GPs engage to enroll 8-12 patients, with requests for participation made to all patients meeting inclusion criteria. Eligible patients are:

* Postmenopausal women
* With (newly) diagnosis of osteoporosis (BMD T-scores ≤ -2.5) OR eligible for anti-osteoporosis treatment because of (previous) fragility fracture after the age of 50 years
* Without terminal illness
* Who are able to speak and understand Dutch
* Who are able to give informed consent Patient eligibility will be judged and patients included by the participating GPs.

Due to current challenges in osteoporosis management, including the unavailability of a locally applicable univocal treatment guideline for PC osteoporosis management, the limited awareness of GPs[2] resulting in underdiagnosis[1, 24] and the treatment gap[1, 24, 25], a guideline for the PC management of PO, hereafter the 'treatment guideline', was developed to improve awareness and case-finding and to standardise treatment and follow-up.

The researchers performed a thorough literature search and consolidated the information from the most recent osteoporosis management guidelines and strategies from several western countries [26-32]. This was subsequently discussed with a scientific steering committee (SSC) representing medical stakeholders in osteoporosis care and adapted to Belgium reimbursement criteria for dual X-ray absorptiometry (DXA) and pharmacological treatment. Because no consensus could be reached during the first SSC assembly, the results were presented to two external osteoporosis experts, and their recommendations incorporated, followed by re-presentation to the SSC. This process was repeated until final consensus.

Bone Friendly Diet Current nutritional advice for women with PO is often directed towards sufficient calcium and vitamin D intake and limited alcohol use[26, 27, 29], despite emerging evidence for other nutritional components impacting BMD[30, 33, 34] or fracture risk[4] and growing scientific conjecture of the relationship between osteoporosis and chronic subclinical inflammation[5, 35] which might be modified through diet[11]. These associations highlight the need for a broader nutritional approach, which has shown to be effective in the management of other chronic diseases[36-38], and in risk reduction, disease prevention and health promotion[39, 40].

Based on the evidence for the roles of Vitamin D and calcium in bone mineralisation[1, 4, 33, 41] and other health factors[37, 40] and the beneficial effects of a Mediterranean-like dietary pattern on diseases and health risks[40, 42, 43], including osteoporosis[11, 34, 44], a Mediterranean diet-based approach has been developed with contributions of registered dietitians to result in the Bone Friendly Diet which is incorporated in the patient education brochure.

Patient information brochure (PIB) A literature search on effective fracture prevention measures was performed. Non-pharmacological aspects of treatment incorporated in the brochure are exercise, nutrition, sunlight exposure, limiting alcohol intake and smoking cessation. To improve patient-friendliness, knowledge on exercise and nutrition were discussed with physiotherapists and dietitians respectively, and underlying principles translated into practical recommendations. For the pharmacological treatment, a chapter is dedicated to the importance of treatment adherence, and scientific information on most frequent incorrect assumptions of anti-resorptive treatment were incorporated. Together with general information on osteoporosis, the information and recommendations is summarised in the PIB.

Nurse education information To support the nurse-educators in their role, an educational map was developed based on the PIB with additional information on epidemiology and pathophysiology, and material to support self-management in patients with chronic disease.

Clinical phase:

Physician level interventions:

Prior to patient inclusion, a researcher will conduct a 45-minute educational session with each participating GP in the doctor's office on the clinical aspects and the multidisciplinary management of PO. Each GP will receive a plasticised A3 version of the treatment guideline for use during clinical practice. Prior to the education, the GPs will complete a survey on osteoporosis management.

Three months after patient enrolment, the GPs will participate in an interactive 2-hour postgraduate education focusing on osteoporosis management, integrated care (IC) for chronic disease and the role of (nurse-)educators in chronic disease management. They will evaluate the treatment guideline by means of an adapted version of the AGREE II [45] questionnaire, to further improve the implementation feasibility. This session will be led by a professor in family medicine specialised in PC organisation and chronic disease management and a professor in rheumatology specialised in bone metabolism, densitometry and osteoporosis.

During the study period, GPs will be supported by a nurse-educator and pharmacists who will have received training in osteoporosis care. They will be encouraged to collaborate with physiotherapists and dietitians for additional support in the management and maintenance of patients' lifestyle changes by means of referral indicators incorporated in the treatment guideline to facilitate collaborative practices.

The nurse-educator will provide assistance to the GPs through:

educating patients with osteoporosis on non- and pharmacological aspects of fracture prevention and supporting their self-management detailed reporting of patient's idea's, needs, concerns, difficulties and obstacles related to (non-)pharmacological treatment adherence supporting collaborative practices between and referral to other PC stakeholders after assessing patients and their living environments and enhancing patient-physician communication by supporting patients in addressing difficulties in osteoporosis management in consultation with their GP and by directly relating important issues to GPs after patient assessment

The pharmacist will provide assistance to the GP through:

reminding patients who have not collected their medications and motivating them to attend new GP consultation to obtain required prescriptions and enhancing patient-physician communication via a standardised referral letter for the pharmacists, that relates difficulties with treatment adherence, the lack of vitamin D and/or calcium in patients' medication lists and/or medication interactions.

The physiotherapist will provide assistance to the GPs through:

performing fall risk assessments in patients with decreased mobility, gait disturbances or other relevant limitations designing personalised exercise programmes for patients to incorporate in their daily routines supervising patients' exercises during physiotherapist consultations and addressing patients' fear of falling.

The dietitian will provide assistance to the GP through:

performing dietary assessments in patients not meeting daily caloric and/or nutritional requirements or suffering from multiple conditions restricting food choices, and providing meal plans and anti-inflammatory food choices for patients with limited intake of qualitative food with regard to calories and nutritional value.

Patient-level intervention:

Patients will receive an IOC-programme package including:

the PIB support from a patient-dedicated, trained nurse-educator specialised in osteoporose care and self-management support, consisting of a home-based 60-90 minute education and support session after study enrolment, with the emphasis on the importance of treatment adherence and lifestyle changes to safeguard BMD. This will be done in a patient-centred manner by addressing all life areas using the 'Zelf-management web' and the setting of personal goals (e.g. dietary changes, treatment adherence improvement, exercise programme implementation) person-tailored telephone follow-up on treatment adherence and the integration of disease management in daily living, beginning 14 days after the educational session and focusing on enhancing intrinsic motivation and implementing disease management in daily living, based on patient preferences a follow-up home-based evaluation session 3 months after the first session to assess progress towards personal goals, set new goals or address barriers preventing goal achievement and support from their pharmacist, consisting of a counseling interview on correct medication administration and intake of osteoporosis medication, the use of calcium and vitamin D, tackling medication side effects and lifestyle practices for bone health informational brochures developed by federal general association of pharmacists(APB) on Osteoporosis, the use of bisphosphonates and calcium/vitamin D or the use of denosumab and calcium/vitamin D - depending on the patients' medications and a referral letter with which the pharmacist can inform the patient's GP on topics discussed (e.g. side effects, medication interactions) and propose solutions to support patients in addressing barriers to treatment adherence.

support from a physiotherapist, consisting of fall risk assessment when indicated due to factors such as limited mobility, gait disturbance or other factors affecting fall risk personalised exercises and addressing fear of falling and fall-efficacy, and supervision during exercises and education on which exercises are safe to perform at home, and support from a dietitian, consisting of specialised education on dietary decisions in cases of multiple conditions requiring nutritional adaptations or restricting food choices, and help in achieving and maintaining a healthy body weight

Pharmacist-level intervention All pharmacists located in GRG will be invited to a postgraduate education prior to patient inclusion. During this 2-hour session, they will receive education on osteoporosis and barriers to treatment adherence, and the roles of the pharmacist in addressing and supporting treatment adherence and communication with patients, family members and GPs. This will be provided in collaboration with the APB and the East-Flanders' association of pharmacists(KOVAG) , and led by a physician and a pharmacist from the APB. The pharmacists will receive patient materials and personal supportive information on osteoporosis and the counseling interview.

As patients have free choice of pharmacists, and we expect only a fraction of the 240 pharmacists in GRG to attend the postgraduate training, all pharmacists in the intervention region will be informed about the project and their role by letter. They will receive the educational material and will be invited to watch the postgraduate training online by means of PowerPoint presentations with voice-over that will be provided on the APB website.

Physiotherapist-level intervention All physiotherapists in the GRG will be invited to a postgraduate education prior to patient inclusion. During this 4.5-hour session, they will receive education on the basic principles and practical management of osteoporosis in physiotherapy, dealing with patients' fear of falling and supporting patients' adherence to exercise and rehabilitation programmes. This education will include lectures from a physician, a university physiotherapy instructor and a PhD researcher. Topics that will be addressed are BMD and PO, and evidence from the literature on the effects of exercise on BMD and fear of falling (physician), practical exercises for BMD maintenance (physiotherapy instructor) and improvement and stimulation of patients' intrinsic motivation to initiate and adhere to behavioural changes (PhD researcher).

Outcomes To measure the impact of and IOC-programme on patients, healthcare providers and society, outcomes will be measured using surveys, data from the InterMutualistisch Agentschap (IMA) and data retrieved from the electronic medical record (EMR).

Primary outcome:

The primary research outcome is the patient's medication possession ratio (MPR) for all antiresorptive treatments during the 12-month study period, starting 12 months prior to the inclusion day and lasting 3 months thereafter, for full coverage of the study period. Patient data on MPR for anti-resorptive treatment will be collected from the IMA-database in a pseudomized manner and a between-group comparison will be performed.

Secondary outcomes:

Secondary outcomes are measured in GPs and patients. Over an 18-month period, the following GP outcomes will be measured in both study arms:

identification failure rate; defined as the proportion of patients eligible for DXA in whom no DXA was performed correct use of the treatment guideline; defined as osteoporosis management in patients who gave informed consent proportion of patients in whom PO is managed appropriately; defined as the proportion of patients eligible for anti-resorptive treatment in whom pharmacological treatment was initiated and/or continued during the study time period correct EMR registration of osteoporosis and -related outcomes; defined as the correct EMR registration of osteoporosis as diagnosis, outcomes of technical investigations (laboratory results, X-ray, DXA, …) and pharmacological treatment for osteoporosis intensity of collaborative practices; defined as the proportion of patients referred to caregivers from the primary or secondary multidisciplinary bone health team by the GP and knowledge of osteoporosis management and treatment

During a 12-month period, the following patient outcomes will be measured using self-reported methods:

health-related competencies in patients (health literacy and self-management efficacy) treatment adherence nutrition medication intake intensity of IOC patient satisfaction with osteoporosis care patient HRQoL and ADL and use of social and healthcare services Economic evaluation

A cost-effectiveness analysis (CEA) from a healthcare payer perspective will be performed with respect to the current modelling guideline in osteoporosis[46]. Cost-effectiveness of IOC will be assessed at a treshold of €40,000 per QALY gained, based on Belgium gross domestic product (GDP)[47] as recommended by the WHO[48]. An age-dependent state-transition model will be used to assess incremental costs, expected QALYs and expected fracture risk after the implementation of IOC compared to CAU. A cycle-length of 1 year and time horizon of 10 years will be applied, in accordance with the 10-year fracture probabilities as calculated with FRAX® and maximum recommended treatment length with bisphosphonates[49]. Fracture risk probabilities at baseline will be calculated with data obtained from both study groups while fracture risk reduction (FRR) for the different therapeutic regimens will be obtained from the literature. Real-world FRR, which also accounts for adherence, will be calculated using study's MPR-data, thereby stratifying adherence into "high" (MPR >80%), "moderate" (50% ≤ MPR ≤ 80%) and "low" (MPR <50%)[50]. Transition probabilities for each state will be obtained from the literature and adjusted for therapeutic regimen and MPR-category.

In both study arms, costs of osteoporosis care will be calculated. For the IOC-group, these include a yearly GP visit, the cost of anti-resorptive treatment multiplied with the MPR, the cost of a 5-yearly DXA, 2 2-hourly visits from a nurse-educator annually and a yearly pharmacist counseling interview. Resource use data collected within the study will be used to calculate average accompanying costs. In the CAU-group, a similar calculation will be conducted, leaving out costs for a nurse-educator and annual pharmacist counseling interview. Cost per QALY gained will be calculated using the Incremental cost-effectiveness ratio (ICER):

ICER = (Cost(IOC)-Cost(CAU))/(QALY(IOC)-QALY(CAU)) Based on the KCE (Belgian Health Care Knowledge Centre) guidelines for health-economic evaluations in Belgium, future costs will be discounted at 3% and future QALYs at 1.5%[51].

ELIGIBILITY:
Inclusion Criteria:

* Patients Postmenopausal women with osteoporosis Non-institutionalized Able to give informed consent
* Family physicians All family physicians willing to participate

Exclusion Criteria:

* Patients Suffering from a terminal illness
* Family physicians No exclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on postmenopausal status
Study Population: Family physicians and their non-institutionalized postmenopausal patients with osteoporosis (yes or not newly diagnosed) who are able to give informed consent for participation within the study.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Medication Possession Ratio (MPR) | 12 months
  Medication Possession Ratio is the sum of the days' supply for all fills of a given drug in a particular time period, divided by the number of days in the time period.

SECONDARY OUTCOMES:
Identification Failure rate | 18 months
  Percentage of women of where not offered DXA despite there eligibility based on risk factors, previous fragility fracture or clinical suspicion of a vertebral fracture
Correct use of the osteoporosis treatment guideline | 18 months
  Percentage of family physicians who implement the osteoporosis treatment guideline in the correct way in patients accepting treatment offered. This is defined as screening with DXA, treatment and follow-up as stated in the treatment guideline.
Proportion of patients treated correctly | 18 months
  The proportion of patients who where eligible for screening and/or treatment that were managed in the correct way as stated in the treatment protocol.
Percentage of family physicians who correctly register osteoporosis management in the EMR | 18 months
  The percentage of family physicians that correctly registers in the EMR the reimbursed fraction of the management and treatment of postmenopausal osteoporosis patients.
Intensity of collaborative practices | 18 months
  The proportion of patients that is referred to one or more professional caregivers for the management of postmenopausal osteoporosis.
Knowledge of osteoporosis management and treatment | 18 months
  Average score on an osteoporosis knowledge test
Health-related competencies | 12 months
  The proportion of patients that has sufficient health-literacy and self-management efficacy for osteoporosis management
Self-reported treatment adherence | 12 months
  The proportion of patients that reports that reports >80% treatment adherence for anti-osteoporotic medication
Self-reported nutritional intake | 12 months
  the proportion of patients that meets daily nutritional requirements as recommended by the healthy bone diet
Self-reported medication intake | 12 months
  The proportion of patients correctly reporting their osteoporosis medication, calcium and Vitamin D supplements
Intensity of integrated osteoporosis care | 12 months
  The proportion of patients that used one or more aspects of an integrative approach by consulting other caregivers and the intensity with which they did it.
Patient satisfaction with osteoporosis care | 12 months
  Proportion of patients that was satisfied with the care that was provided with the different caregivers they consulted for their osteoporosis care
Patient Health Related Quality of Life (HRQoL) | 12 months
  Evolution of HRQoL presented as QALY's
Patient functional independence | 12 months
  Evolution of functional independence expressed as activities of daily living (ADL) patients
Resource use | 12 months
  The identification of, duration of and frequency with which social and healthcare services used by patients

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Borgermans, PhD, Study Chair — University Ghent
Locations (1):
- Family physician doctor's offices, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verdonck C, Annemans L, Goemaere S, Lapauw B, Goderis G, Balligand E, Doom MP, Perkisas S, Borgermans L. The effectiveness and cost-effectiveness of an integrated osteoporosis care programme for postmenopausal women in Flanders: study protocol of a quasi-experimental controlled design. Arch Osteoporos. 2020 Jul 22;15(1):107. doi: 10.1007/s11657-020-00776-7. PMID 32700114